CLINICAL TRIAL: NCT02774369
Title: Improving Sleep Among Cancer Patients: Comparison Between Physical Activity and Self-administered Cognitive-behavioral Therapy (CBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Josée Savard, Researcher, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-933, A12-04-933
Record Dates: First submitted 2016-05-04; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Cancer; Insomnia
Keywords: cancer; insomnia; sleep; physical exercise; aerobic; cognitive-behavioral therapy; self-help; RCT
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical exercise (Experimental): A 6-week individualised, aerobic intervention program elaborated by a kinesiologist following a complete assessment of the individual's physical condition.
  Interventions: Behavioral: Physical exercise
- Cognitive-behavioral therapy (Active Comparator): A 6-week self-administered cognitive-behavioral therapy for insomnia composed of a 60-min video (DVD format) and 6 booklets.
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Physical exercise — Individualized aerobic intervention program
  Arms: Physical exercise
Behavioral: Cognitive-behavioral therapy — Psychological intervention combining behavioral, cognitive, and educational strategies
  Other Names: CBT
  Arms: Cognitive-behavioral therapy

SUMMARY:
It has been suggested that the practice of physical exercise can improve sleep, but few studies have investigated this issue in the context of cancer, despite the proven benefits of exercise in this population. This randomized-controlled trial (RCT) aimed to compare the efficacy of an aerobic intervention program to that of a self-administered cognitive-behavioral therapy (CBT) to improve sleep of cancer patients. Forty-one men and women with insomnia symptoms and treated within 6 months for a non-metastatic cancer participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of non-metastatic cancer
* adjuvant treatments completed within the past 6 months
* insomnia symptoms as defined by a score ≥ 8 on the Insomnia Severity Index
* practicing less than 90 minutes of physical exercise per week
* able to readily read and understand French
* available during a consecutive 6-week period to complete the intervention
* written permission from physician to engage in a physical exercise program

Exclusion Criteria:

* severe cognitive impairments (e.g., diagnosis of Parkinson disease)
* severe psychiatric disorder (e.g., severe major depression)
* diagnosis of a sleep disorder other than insomnia (e.g., obstructive sleep apnea)
* any contraindication for the practice of physical exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index total score | Pre-tx (at recruitment, T1); Post-tx (6 weeks after, T2), 3-month FU (T3), 6-month FU (T4)
  A 7-item questionnaire evaluating the perceived severity of sleep difficulties. The total score is the main outcome (ranging from 0 to 28).

SECONDARY OUTCOMES:
Change in sleep efficiency (SE) index (%) | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4)
  total sleep time/total time spent in bed X 100 - from sleep diary
Change in sleep onset latency (SOL) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4)
  time to sleep after lights out - from sleep diary
Change in wake after sleep onset (WASO) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4)
  summation of nocturnal awakenings - from sleep diary
Change in total sleep time (TST) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4)
  time in bed minus total wake time - from sleep diary
Change in Fatigue Symptom Inventory total score | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4)
  A 15-item questionnaire measuring perceived fatigue. The total score ranges from 15 to 75.
Change in Hospital Anxiety and Depression Scale | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4)
  A 14-item questionnaire comprising 7 items assessing depression (HADS-D) and 7 items assessing anxiety (HADS-A). Scores obtained for each subscale range from 0 to 21.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Mercier J, Ivers H, Savard J. A non-inferiority randomized controlled trial comparing a home-based aerobic exercise program to a self-administered cognitive-behavioral therapy for insomnia in cancer patients. Sleep. 2018 Oct 1;41(10). doi: 10.1093/sleep/zsy149. PMID 30053196